CLINICAL TRIAL: NCT02856776
Title: RCT Double Blinded Evaluation of Changes in Gene Expression, Metabolomic, Microbiome, and Calcium Metabolism in Response to Varied Vitamin D Dosages in Adults Who Are Vitamin D Insufficient
Brief Title: Gene Expression, Metabolomic, Microbiome, and Calcium Metabolism in Response to Varied Vitamin D Dosages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Pure North S'Energy Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: H-35506
Record Dates: First submitted 2016-07-28; First posted 2016-08-05 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Vitamin D Insufficiency
Keywords: Vitamin D; Metabolomics; Microbiota; Gene Expression
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1: 600 IU vitamin D (Experimental): Subject will receive 600 IUs of vitamin D3/day for 24 weeks.
  Interventions: Dietary Supplement: Vitamin D3
- Arm 2: 4,000 IU vitamin D (Experimental): Subject will receive 4,000 IUs of vitamin D3/day for 24 weeks
  Interventions: Dietary Supplement: Vitamin D3
- Arm 3: 10,000 IU vitamin D (Experimental): Subjet will receive 10,000 IUs of vitamin D3/day for 24 weeks
  Interventions: Dietary Supplement: Vitamin D3
- Arm 4: Mixed vitamin D dosages (Experimental): Subject will receive 600 IUs of vitamin D3/day for the first 8 weeks, 4,000 IUs of vitamin D3/day for the next 8 weeks, and 10,000 IUs of vitamin D3/day for the final 8 weeks.
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Vitamin D provided in capsule form

SUMMARY:
There continues to be debate as to how much vitamin D an adult requires to be vitamin D sufficient. A multitude of association studies have suggested that improving serum 25(OH)D >30 ng/mL may reduce risk of many chronic illnesses and improve immune function. The aim of this study is to define dynamic changes in PTH, broad gene expression in circulating immune cells, metabolomics, and microbiome profile in response to varying doses of vitamin D supplementation.

DETAILED DESCRIPTION:
Vitamin D requires two metabolic conversions, 25-hydroxylation in the liver and 1α-hydroxylation in the kidney, before its hormonal form, 1,25-dihydroxyvitamin D [1,25(OH)2D], can bind to the vitamin D receptor (VDR) to modulate gene transcription. The VDR is present in a wide variety of cells and tissues and 1,25(OH)2D via its receptor directly or indirectly have been reported to have effects on cell cycling and proliferation, differentiation, apoptosis and the production of cathelicidin, renin and insulin. It is estimated that VDR activation may regulate directly and/or indirectly the expression of a very large number of genes (0.5-5% of the total human genome i.e., 100-1250 genes). Early microarray studies performed in squamous carcinoma and osteoblasts cells revealed that 1,25(OH)2D3 regulated the expression of numerous genes including those implicated in immune function . Although there have been numerous observations of vitamin D deficiency and its links to chronic diseases, a study on how a person's vitamin D status and improvement with vitamin D supplementation affects genomic expression in vivo in humans had not been reported until recently when we observed in a small pilot study that supplementation of healthy adults with vitamin D significantly affected the expression of 291 genes that have been linked to more than 80 different metabolic pathways. This small randomized controlled double blind study funded by our CTSI and registered in Clinical Trials.gov (NCT01696409) included 2 groups. Group 1 received 400 IUs of vitamin D3 (400 IUs at the time of the study in 2010 was before the IOM released its new recommendations) and was considered the control group and group 2 received 2000 IUs of vitamin D3 daily for 2 months during the winter. Comparing gene expression in these two groups (deficient vs. insufficient or sufficient) led us to study the effect of vitamin D status as well as vitamin D supplementation on genome-wide gene expression. To explore gene-expression relationships between and within the 400 IU and 2000 IU groups, principal component analysis (PCA) was performed. We observed the same trend in gene expression in the subjects who received 400 and 2000 IUs vitamin D3. There was however a trend for a larger change in the expression of these genes for the group who received 2000 IUs vitamin D3/d compared to the group who received 400 IUs vitamin D3/d. Regarding all participants, with false discovery rate (FDR) < 0.1, and a 1.5 fold change, 291 genes were found to have a statistically significant difference in expression from baseline to follow-up after vitamin D3 supplementation. There was at least a 1.5 fold inhibition of 82 genes (top ~30% of the heat map) whose expression was dramatically reduced and at least a 1.5 fold induction of 209 genes (bottom ~70% of the heat map) whose expression was significantly increased after supplementation with either 400 or 2000 IU of vitamin D3 for 2 months. For verification that genes that we observed to have their expression affected by vitamin D supplementation did occur expression changes were evaluated by real-time PCR for four genes including CD83, TNFAIP3, KLF10 and SBDS. The gene expression changes were concordant with those observed by the microarray analysis.

This subgroup analysis of the baseline gene expression for the 291 genes in the vitamin D deficient group compared to the vitamin D insufficient/sufficient group revealed that, expression of 66 genes were significantly different between the two groups (p<0.01 and fold change>1.5). There was at least a 1.5 fold increase in gene expression (brown-orange) of 14 genes and at least a 1.5 fold decrease in the expression (yellow-white) of 52 genes in the vitamin D deficient adults compared to those who were vitamin D insufficient or sufficient at baseline. After vitamin D3 supplementation gene expression in the vitamin D deficient group was similar to vitamin D insufficient/sufficient group. To learn which of these genes affected by vitamin D3 supplementation contained VDR binding domains near the transcriptional start site (TSS), we performed a VDRE analysis. Of the 66 genes that were influenced by at least 1.5 fold in their expression by the baseline serum 25(OH)D concentration,17 of these genes that were significantly changed after vitamin D3 supplementation in both deficient and insufficient/sufficient groups (p<0.01) were selected for VDRE analysis. We found at least one candidate VDRE in the upstream region within 30 kb of the TSS in these 17 genes. For example, the candidate VDRE in coatomer protein complex, subunit beta 2 (COPB2), a gene that was stimulated at least 1.5 fold by vitamin D3 supplementation, had two hexameric binding motifs associated with the VDRE. Twelve housekeeping genes served as negative controls. There were no sequences of candidate VDREs in 100 kb upstream of TSS of these housekeeping genes and the expression of these housekeeping genes after vitamin D3 supplementation was not changed.

VDR is present in a wide variety of cells and tissues, in particular they are prominent on cells involved in innate and adaptive immunity; especially CD8+ T lymphocytes.These immune cells are found throughout the body including parts of the digestive tract. In particular, the upper GI tract (including the pyloric antrum and duodenum) has the greatest concentration of CD8+ T cells relative to the rest of the GI tract. Studies have found that those who increase their vitamin D intake have a reduction in opportunistic pathogens and an increase in gut microbiome. Through the action of vitamin D on CD8+ T cells, there is an increase immune response against gammaproteobacteria which allows the gut microbiome to flourish. This study found that although the upper GI tract generated the greatest change in microbiome secondary to vitamin D supplementation, the rest of the GI tract and stool also displayed a change. Gut microbiome is important for general health maintenance. For example, changes in gut microbiota have been associated with early onset of Type 2 - Diabetes Mellitus (T2DM). Thus, it is possible to understand the prevalence of VDR expression on immune cells in an individual by observing the microbiota in the gut/stool.

The objective of this proposed project will be to expand on these preliminary data in a well-defined group of healthy adults ages 18-50 years with a BMI <30 kg/m2 who are vitamin D insufficient with a 25(OH)D of < 29 ng/mL

There continues to be debate as to how much vitamin D an adult requires to be vitamin D sufficient. A multitude of association studies have suggested that improving serum 25(OH)D >30 ng/mL may reduce risk of many chronic illnesses and improve immune function. 1,25-dihydroxyvitamin D3 [1,25(OH)2D] may regulate at least 2000 genes. Our recent pilot study evaluating the effect of vitamin D status and vitamin D supplementation on broad gene expression revealed as many as 291 genes are influenced by vitamin D3 supplementation.

Aim: Define Dynamic Changes in PTH, Broad Gene Expression in Circulating Immune Cells, metabolomics, and microbiome profile in Response to Varying Doses of Vitamin D Supplementation.

The hypothesis that will be tested is that as serum 25(OH)D levels increase as a result of vitamin D supplementation there will be a gradual decline in PTH levels. Furthermore we expect that there will continue to be alterations in gene expression, metabolomic protein levels and in the gut microbiome when the dose is increased to 10,000 IUs daily whereas the PTH levels will plateau at a dose of 4000 IUs daily and remain the same when the dose is escalated to 10,000 IUs daily.

This study will last 24 weeks and blood, urine, and stool samples will be obtained at baseline and at 8 week intervals to evaluate the time course for the changes in 25(OH)D, PTH levels, gene expression, and determine if these changes remain constant or are continuing to change after vitamin D supplementation. We will conduct a metabolomics profile in blood and urine as well as determine if there are any microbiome changes in the stool as previously described. In addition, one arm of the study will include a group who will receive 600 IUs for the first 8 weeks followed by 4000 IUs for the next 8 weeks followed by 10,000 IUs of vitamin D3 for the final 8 weeks to determine whether continued increase in vitamin D intake in the same adult will continue not only to alter gene expression, metabolomics activity, and microbiome changes, but also influence PTH levels. Although the IOM's UL for vitamin D for adults is 4000 IU/D they and the Endocrine Society recognized that up to 10,000 IUs/D was safe in healthy adults for up to 5 months. In addition a recent study reported that adults taking up to 20,000 IUs/D for at least one year never raised their blood level above 250 nmol/L i.e. 100 ng/mL which is considered by the IOM, Endocrine Society and many reference laboratories to be the upper limit of normal. Results from this study should provide a new insight as to how much vitamin D a healthy adult requires to maximize their calcium and bone metabolism and expression of genes related to the immune system and other biologic pathways in the blood, urine, and stool.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female adults
2. Age 18-50 years
3. BMI <30
4. 25-hydroxyvitamin D < 29 ng/mL
5. No medications or disorders that would affect vitamin D metabolism
6. Women must be on birth control and not pregnant based on a negative pregnancy test at baseline
7. Ability and willingness to give informed consent and comply with protocol requirements

Exclusion Criteria:

1. Ongoing treatment with pharmacologic doses of vitamin D, vitamin D metabolites or analogues
2. Pregnancy
3. History of elevated serum calcium (>10.6 mg%); that is corrected for albumin concentration
4. Chronic hepatic or renal failure
5. Supplementation with over the counter formulations of vitamin D2 or vitamin D3
6. Subjects with a history of an adverse reaction to orally administered vitamin D.
7. Subjects who are taking oral Dilantin or glucocorticoids.
8. History of intestinal malabsorption (i.e. cystic fibrosis, fat malabsorption syndrome, Crohn's Disease, gastric bypass surgery).
9. Inability to give informed consent
10. Vacation plans to warmer climates (Florida, Southern CA, tropics) during study participation
11. Subjects with any other condition which in the Investigator's judgment would make the patient unsuitable for inclusion in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-08-06 (Actual)

PRIMARY OUTCOMES:
Change in Gene Expression in circulating immune cells | Baseline and 24 weeks
  Change in gene expression of VDR receptors located on circulating immune cells.
Change in Metabolomic profile - Carbohydrates | Baseline and 24 weeks
  Change in carbohydrate profile of blood and urine i.e. Glucose (mg/dL)
Change in Stool microbiome | Baseline and 24 weeks
  Change in microbiota of the stool
Change in Metabolomic profile - Amino Acids | Baseline and 24 weeks
  Change in amino acid profile of blood and urine i.e. Lysine (mg/dL)
Change in Metabolomic profile - Small Peptides | Baseline and 24 weeks
  Change in small peptide profile of blood and urine i.e. stearic acid (mg/dL)
Change in Metabolomic profile - Lipids | Baseline and 24 weeks
  Change in lipid profile of blood and urine i.e. cholesterol (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Holick, MD,PhD, Principal Investigator — Boston University
Locations (1):
- Boston University Medical Campus, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No